CLINICAL TRIAL: NCT02632461
Title: The Dietary Intervention Examining Tracking With Mobile Devices Study
Brief Title: Dietary Intervention Examining Tracking With Mobile Devices
Acronym: DIETMobile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Brie Turner-McGrievy, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00049756
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Obesity
Keywords: Diet; Weight Loss; Tracking; Calories
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Podcast (+Bite Counter) (Experimental): Participants in this group will receive podcasts twice weekly in conjunction with using a wearable wrist device called a Bite Counter. The Bite Counter tracks the number of bites/calories per bite. (Podcasts plus Bite Counter)
  Interventions: Behavioral: Podcasts; Behavioral: Bite Counter
- Podcast (+Mobile App) (Active Comparator): Participants in this group will receive podcasts twice weekly in conjunction with using a mobile application to track their diet. (Podcasts plus Mobile Diet Application)
  Interventions: Behavioral: Podcasts; Behavioral: Mobile Diet Application

INTERVENTIONS:
Behavioral: Podcasts — Participants will receive twice weekly podcasts that will cover topics related to weight loss.
Behavioral: Mobile Diet Application — Participants will use a mobile application on their smartphone to track their diet.
  Arms: Podcast (+Mobile App)
Behavioral: Bite Counter — Participants will use a wrist-worn Bite Counter to track the number of bites in their diet per day.
  Arms: Podcast (+Bite Counter)

SUMMARY:
The purpose of the study is to test the effectiveness of two different weight loss interventions. Both of these interventions will provide weight loss information through twice weekly audio podcasts. In addition to the podcasts, participants will be asked to track their diet using either a wearable device on their wrist or through an app on their smartphone.

DETAILED DESCRIPTION:
This study will last approximately 6 months. Participants will attend one 1-hour orientation meeting at the beginning of the study and a 2-hour baseline assessment and training meeting. Additional assessments will be conducted at 3 months and 6 months. Weekly questionnaires will be administered. Everyone in the study will be asked to listen to 2 podcasts per week. Each of the podcasts will take about 15 - 20 minutes to listen to and so participants should expect to spend 30 - 40 minutes each week listening to podcasts. Participants will also be randomized to either track diet with an app on their smartphone or using a device they wear on their wrist. Each week, participants will be sent an email as a reminder on how to use their diet tracking device. They will also be encouraged to monitor their exercise and body weight.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18-65 years old
* Own and use a smartphone and/or a tablet with a data plan
* BMI must be between 25-49.9 kg/m2
* Must be willing to reduce caloric intake and increase physical activity
* Not currently participating in a weight loss study in a weight loss study that involved podcasts

Exclusion Criteria:

* Over the age of 65 years old
* Currently participating in a weight loss program
* Has lost more than 10 pounds in the past 6 months
* Diagnosed with stroke or heart attack
* Diagnosed with diabetes that is controlled using medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in body weight as assessed by digital scale | 6 months
  Change in body weight from baseline to 6 months as assessed by digital scale.

CONTACTS AND LOCATIONS:
Overall Officials: Brie Turner-McGrievy, Principal Investigator — University of South Carolina School of Public Health
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Turner-McGrievy GM, Dunn CG, Wilcox S, Boutte AK, Hutto B, Hoover A, Muth E. Defining Adherence to Mobile Dietary Self-Monitoring and Assessing Tracking Over Time: Tracking at Least Two Eating Occasions per Day Is Best Marker of Adherence within Two Different Mobile Health Randomized Weight Loss Interventions. J Acad Nutr Diet. 2019 Sep;119(9):1516-1524. doi: 10.1016/j.jand.2019.03.012. Epub 2019 May 30. PMID 31155473
- [Derived] Turner-McGrievy GM, Wilcox S, Boutte A, Hutto BE, Singletary C, Muth ER, Hoover AW. The Dietary Intervention to Enhance Tracking with Mobile Devices (DIET Mobile) Study: A 6-Month Randomized Weight Loss Trial. Obesity (Silver Spring). 2017 Aug;25(8):1336-1342. doi: 10.1002/oby.21889. Epub 2017 Jun 10. PMID 28600833